CLINICAL TRIAL: NCT03112018
Title: Strengthening Intrapartum and Immediate Newborn Care to Reduce Morbidity and Mortality of Preterm Infants in Health Facilities in Migori County, Kenya and Busoga Region, Uganda: an Implementation Science RCT
Brief Title: Strengthening Facility-based Intrapartum/Immediate Newborn Care to Reduce Mortality of Preterm Infants in Migori County, Kenya and Busoga Region, Uganda
Acronym: PTBi-KE-UG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Makerere University (Other); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dilys Walker, Principal Investigator, Preterm Birth Initiative East Africa; University of California, San Francisco, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A123218-K/U
Record Dates: First submitted 2016-12-19; First posted 2017-04-13 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Pregnancy Complications; Preterm Labor; PreTerm Birth; Stillbirth; Low Birth Weight
Keywords: premature birth; neonatal mortality; premature infant
MeSH Terms: conditions — Pregnancy Complications; Obstetric Labor, Premature; Premature Birth; Stillbirth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator): * Data strengthening
  * modified Safe Childbirth Checklist (mSCC) implementation
  Interventions: Behavioral: data strengthening; Behavioral: modified Safe childbirth checklist - control
- Enhanced care (intervention) (Experimental): * Data strengthening
  * modified Safe Childbirth Checklist (mSCC) implementation
  * Health provider training (PRONTO)
  * Quality Improvement (QI) Cycles
  Interventions: Behavioral: data strengthening; Behavioral: modified Safe childbirth checklist - enhanced; Behavioral: PRONTO training; Behavioral: QI cycles

INTERVENTIONS:
Behavioral: data strengthening — Data strengthening: initial training, monthly data collection and feedback on data quality, access to dashboards, periodic Data Quality Assessments
Behavioral: modified Safe childbirth checklist - control — modified Safe Childbirth Checklist (mSCC) implementation: provision of the mSCC to facilities, limited feedback and mentoring on its use
  Arms: Standard care
Behavioral: modified Safe childbirth checklist - enhanced — modified Safe Childbirth Checklist (mSCC) implementation: provision of the mSCC to facilities, ongoing intensive feedback and mentoring on its use
  Arms: Enhanced care (intervention)
Behavioral: PRONTO training — Health provider training (PRONTO): initial 2-days modular training followed by a 6-week mentoring sessions (Kenya) or periodic modular refreshers and supplemental mentoring (Uganda), each over a 9-12 month period
  Arms: Enhanced care (intervention)
Behavioral: QI cycles — Quality Improvement Cycles (QI): facility teams performing PDSA cycles with mentoring support and twice annual Learning Collaborative sessions, plus opportunities to apply for small amounts of funds to support change efforts
  Arms: Enhanced care (intervention)

SUMMARY:
The purpose of this study is to determine whether a combination of evidence-based strategies can improve intrapartum and newborn care in facilities to reduce mortality among preterm infants. This will be a cluster randomized implementation science study across 23 facilities in Eastern Uganda and Western Kenya. Selected interventions will be supported in facilities to measure impact during the study period. These interventions are: a) data strengthening and data use activities; b) implementation of a modified WHO Safe Childbirth Checklist with an emphasis on preterm labor and preterm babies; c) simulation-based provider training and mentoring on key existing evidence-based practices to improve newborn outcomes; d) support of Quality Improvement (QI) cycles to identify and resolve facility-specific issues and bottlenecks. A two-stage design will be used where all study facilities will receive some aspects of the intervention initially, namely data strengthening and the modified checklist. Subsequently, the remaining interventions (QI cycles and simulation training of providers) will be rolled out to a randomly selected half of the facilities in the first stage. At a second stage, the remaining half of the facilities will receive the remaining interventions.

DETAILED DESCRIPTION:
The randomized, controlled cluster trial (RCCT) will test whether the study intervention reduces the combined incidence of fresh stillbirth and neonatal mortality by 30% compared with the control group incidence of FSB+NMR. Given a Type I error of 0.05, power=80%, a one-tailed test, a balanced (1 control :1 intervention) sample, and a baseline PTB NMR of 10%, the RCCT requires 1,133 PTBs in each study group. The sample size has been increased by 35% to account for a 25% design effect and a 10% loss to follow-up/missing information, requires 1,530 PTBs in each study group. Secondary outcomes will be assessed using this sample. The study randomized facilities to either the control or intervention group, matched on various characteristics to improve the similarity of the study groups and minimize design effect. This a priori hypothesis is proposed prior to analyzing the intervention period study primary outcome, using the baseline PTB incidence of FSB+NMR, and an effect size previously observed with PRONTO.

This implementation science study includes a package of interventions. Control sites receive only the limited package of data strengthening and implementation of the modified Safe Childbirth Checklist. The randomly selected intervention facilities receive an enhanced package which also includes provider training/mentoring using PRONTO simulation and teamwork training, ongoing clinical mentoring, and support for Quality Improvement cycles (PDSA cycles) using a Model for Improvement framework. More detail about the contents of the intervention is included below.

Data Strengthening Strategies: initial training focused on routinely collected data plus ongoing refreshers and mentorship throughout study duration

* Strengthen the MOH data collection system (birth registries, admission/discharge registries), as well as introduction of expanded documentation to capture preterm birth details
* Perform facility assessment to determine gaps in infrastructure, supplies as well as skills and competencies of providers and data managers to accurately and consistently report routine facility data
* Support facilities to use standardized definitions of indicators currently collected for antenatal and postnatal care
* Support adherence to national guidelines on documentation in the registers and patient charts through training, provision of registers/charts and motivation
* Introduce expanded routine documentation of preterm births including improving the register to capture data on preterm and still births, and implementation of the modified WHO Safe Childbirth Checklist (see below)
* Support periodic data quality assessment cycles
* Create a synchronized online data dashboard repository system representing key indicators on an ongoing basis with selective access for health care providers and national policy makers

WHO Safe Childbirth Checklist modified to address identification of preterm labor and newborn care for preterm babies: initial training plus ongoing refreshers and mentorship throughout study duration

* Introduce expanded routine documentation of preterm births including the piloting and use of a modified WHO Safe Childbirth Checklist (mSCC)
* Introduce and train on use of the mSCC to detect, manage and treat high risk labor/babies
* Collect routine facility data including register reviews (study staff will visit each selected facility at least once per month)
* Conduct periodic audits of the mSCC to determine uptake and completeness, review for phenotyping information, and/or review for additional service indicators on preterm babies

Measures to strengthen, recommended intrapartum, postnatal and neonatal care in facilities through PRONTO simulation-based provider training and mentorship: training of trainers and initial trainings in Kenya and Uganda plus ongoing mentorship in Kenya and modular refreshers in Uganda, throughout study duration

* Improve intrapartum, postnatal and neonatal management by using a customized PRONTO curriculum that includes highly realistic simulation and focused team training to address gaps in emergency obstetric and neonatal response. The training emphasizes lifesaving response during labor, delivery, postnatal and neonatal periods with specific emphasis on the care of preterm babies.
* Initial 2-days modular PRONTO training will be followed by periodic modular refreshers and supplemental mentoring. In Kenya, this involves 6 one-week mentoring sessions led by trained preterm champions over a 9-12 month period. In Uganda, a modular training model with intermittent refresher trainings and two-day clinical mentoring sessions will be offered over a 9-12 month period. Special emphasis will be put on evidence-based practices and the views gathered from Kenya and Uganda stakeholders.
* Promote close follow-up of preterm babies up to 28-days

Measures to strengthen Quality Improvement (QI) cycles: initial training with ongoing mentorship; QI team meetings each week with quarterly cross-facility collaboration workshops throughout study duration

* Develop tools for, introduce and institutionalize QI cycles and regular project monitoring and evaluation
* Reinforcement of accurate and timely documentation in charts and registers in the facilities
* Reinforcement of use of the mSCC, including its use as a data source to track progress of change efforts
* Link system gaps or latent errors uncovered during simulation training and suggested solutions with QI efforts
* Develop and recommend some tools to improve data collection such as for triage, discharge and referral

ELIGIBILITY:
Inclusion Criteria:

* Individuals: Investigators will include in the analysis the birth outcomes of all women accessing delivery care services at selected hospitals with gestational age of > 24 weeks who are either admitted for labor or for hospitalization for another antenatal complication (preeclampsia, chorioamnionitis) or referred to a tertiary hospital. Women will be presenting at either control or intervention sites and their delivery information will be reviewed. For follow-up, the investigators will select women with infants born at greater than 1000 grams and less than 2500 grams, or between 2501 and 2999 grams with documented gestational age less than 37 weeks.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102988 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
all-cause neonatal mortality among preterms/low birth weight newborns | 28-days after facility-based delivery
  To determine the effect of the full package (data strengthening, mSCC, provider training and mentoring using the PRONTO method, QI cycles) on 28-day all-cause mortality rate among low birth weight neonates greater than 1000 grams and less than 2500 grams, and neonates between 2500 and 2999 grams with documented gestational age less than 37 weeks

SECONDARY OUTCOMES:
Data quality of key indicators in facility-based registers | through study completion, an average of 18 months
  Key indicators include gestational age, facility discharge status, preterm birth incidence
Pre-hospital discharge mortality among preterm infants and babies born alive between 500 and 999 grams at birth | at hospital discharge, an average of 1-7 days
28-day mortality among babies born alive between 500 and 999 grams at birth | 28-days after facility-based delivery
Average number of evidence-based practices demonstrated in simulated case videos and live birth observations | Baseline and through study completion, an average of 18 months
  Uptake and appropriate utilization of evidence-based interventions/ Ministry of Health management guidelines measured in PRONTO simulation videos, observed live births and/or mSCC
Prevalence of preterm birth phenotypes in the study sites as measured by chart review and the mSCC | Every year over four years
Facility readiness to handle delivery and newborn complications as measured by a facility assessment tool | Every six months over two years

CONTACTS AND LOCATIONS:
Overall Officials: Dilys Walker, MD, Principal Investigator — University of California, San Francisco; Peter Waiswa, MD, MPH, PhD, Principal Investigator — Makerere University School of Public; Phelgona Otieno, MBChB, MPH, Principal Investigator — Kenya Medical Research Institute
Locations (2):
- Health facilities in Migori County: Rongo, Kehancha, Uriri, Kegonga, Karungu, Tisinye, Isibania, Macalder, Awendo, Ntimaru, Muhuru, Bugumbe, Nyamaraga, Othoro, St. Joseph, St. Camillus, Migori County Referral Hospital, Migori County, Migori County, Kenya
- Health facilities in Busoga Region: Bugiri, Buluba, Iganga, Kamuli Government, Kamuli Mission, Jinja Regional Referral Hospital, Busoga Region, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mandu R, Miller L, Namazzi G, Twum-Danso N, Achola KJA, Cooney I, Butrick E, Santos N, Masavah L, Nyakech A, Kirumbi L, Waiswa P, Walker D. Quality improvement collaboratives as part of a quality improvement intervention package for preterm births at sub-national level in East Africa: a multi-method analysis. BMJ Open Qual. 2023 Dec 21;12(4):e002443. doi: 10.1136/bmjoq-2023-002443. PMID 38135302
- [Derived] Martin-Herz SP, Otieno P, Laanoi GM, Moshi V, Olieng'o Okoth G, Santos N, Walker D. Growth and neurodevelopmental outcomes of preterm and low birth weight infants in rural Kenya: a cross-sectional study. BMJ Open. 2023 Aug 31;13(8):e064678. doi: 10.1136/bmjopen-2022-064678. PMID 37652593
- [Derived] Ghosh R, Otieno P, Butrick E, Santos N, Waiswa P, Walker D; Preterm Birth Initiative Kenya and Uganda Implementation Research Collaborative. Effect of a quality improvement intervention for management of preterm births on outcomes of all births in Kenya and Uganda: A secondary analysis from a facility-based cluster randomized trial. J Glob Health. 2022 Dec 29;12:04073. doi: 10.7189/jogh.12.04073. PMID 36580073
- [Derived] Ghosh R, Santos N, Butrick E, Wanyoro A, Waiswa P, Kim E, Walker D. Stillbirth, neonatal and maternal mortality among caesarean births in Kenya and Uganda: a register-based prospective cohort study. BMJ Open. 2022 Apr 6;12(4):e055904. doi: 10.1136/bmjopen-2021-055904. PMID 35387820
- [Derived] Whaley B, Butrick E, Sales JM, Wanyoro A, Waiswa P, Walker D, Cranmer JN. Using clinical cascades to measure health facilities' obstetric emergency readiness: testing the cascade model using cross-sectional facility data in East Africa. BMJ Open. 2022 Apr 4;12(4):e057954. doi: 10.1136/bmjopen-2021-057954. PMID 35379635
- [Derived] Achola KA, Kajjo D, Santos N, Butrick E, Otare C, Mubiri P, Namazzi G, Merai R, Otieno P, Waiswa P, Walker D. Implementing the WHO Safe Childbirth Checklist modified for preterm birth: lessons learned and experiences from Kenya and Uganda. BMC Health Serv Res. 2022 Mar 3;22(1):294. doi: 10.1186/s12913-022-07650-x. PMID 35241076
- [Derived] Namazzi G, Achola KA, Jenny A, Santos N, Butrick E, Otieno P, Waiswa P, Walker D; Preterm Birth Initiative Kenya & Uganda Implementation Research Collaborative. Implementing an intrapartum package of interventions to improve quality of care to reduce the burden of preterm birth in Kenya and Uganda. Implement Sci Commun. 2021 Jan 28;2(1):10. doi: 10.1186/s43058-021-00109-w. PMID 33509293
- [Derived] Walker D, Otieno P, Butrick E, Namazzi G, Achola K, Merai R, Otare C, Mubiri P, Ghosh R, Santos N, Miller L, Sloan NL, Waiswa P; Preterm Birth Initiative Kenya and Uganda Implementation Research Collaborative. Effect of a quality improvement package for intrapartum and immediate newborn care on fresh stillbirth and neonatal mortality among preterm and low-birthweight babies in Kenya and Uganda: a cluster-randomised facility-based trial. Lancet Glob Health. 2020 Aug;8(8):e1061-e1070. doi: 10.1016/S2214-109X(20)30232-1. PMID 32710862
- [Derived] Otieno P, Waiswa P, Butrick E, Namazzi G, Achola K, Santos N, Keating R, Lester F, Walker D. Strengthening intrapartum and immediate newborn care to reduce morbidity and mortality of preterm infants born in health facilities in Migori County, Kenya and Busoga Region, Uganda: a study protocol for a randomized controlled trial. Trials. 2018 Jun 5;19(1):313. doi: 10.1186/s13063-018-2696-2. PMID 29871696
- See also: PRONTO website — http://prontointernational.org/